CLINICAL TRIAL: NCT03854227
Title: A PHASE 1 STUDY TO EVALUATE THE SAFETY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF ESCALATING DOSES OF PF-06939999 (PRMT5 INHIBITOR) IN PARTICIPANTS WITH ADVANCED OR METASTATIC NON-SMALL CELL LUNG CANCER, HEAD AND NECK SQUAMOUS CELL CARCINOMA, ESOPHAGEAL CANCER, ENDOMETRIAL CANCER, CERVICAL CANCER AND BLADDER CANCER
Brief Title: A Dose Escalation Study Of PF-06939999 In Participants With Advanced Or Metastatic Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study has been terminated based on a strategic evaluation within the current Pfizer oncology portfolio. This decision is not due to any safety concerns or requests from any regulatory authorities.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C3851001
Record Dates: First submitted 2019-02-15; First posted 2019-02-26 (Actual); Results first posted 2025-01-13 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Intervention Model Description: Dose Escalation and Dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose Escalation (Experimental): Participants will receive PF-06939999 orally at escalating doses in 28 day cycles on a continuous basis
  Interventions: Drug: PF-06939999 dose escalation
- Non small cell lung cancer monotherapy (Experimental): Participants will receive PF-06939999 at the recommended Phase 2 dose in 28 day cycles on a continuous basis
  Interventions: Drug: PF-06939999 monotherapy
- Urothelial carcinoma (Experimental): Participants will receive PF-06939999 at the recommended Phase 2 dose in 28 day cycles on a continuous basis
  Interventions: Drug: PF-06939999 monotherapy
- Head and neck squamous cell carcinoma (Experimental): Participants will receive PF-06939999 at the recommended Phase 2 dose in 28 day cycles on a continuous basis
  Interventions: Drug: PF-06939999 monotherapy
- Non small cell lung cancer PF-06939999 plus docetaxel (Experimental): Participants will receive PF-06939999 on a continuous basis in combination with docetaxel
  Interventions: Drug: PF-06939999 in combination with docetaxel
- Non small cell lung cancer dose finding (Experimental): Participants will receive PF-06939999 on a continuous basis at escalating doses in combination with docetaxel
  Interventions: Drug: PF-06939999 in combination with docetaxel

INTERVENTIONS:
Drug: PF-06939999 dose escalation — PF-06939999 orally at escalating doses on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Dose Escalation
Drug: PF-06939999 monotherapy — PF-06939999 at the recommended Phase 2 dose orally on a continuous basis
  Other Names: PRMT5 inhibitor
  Arms: Head and neck squamous cell carcinoma; Non small cell lung cancer monotherapy; Urothelial carcinoma
Drug: PF-06939999 in combination with docetaxel — PF-06939999 orally on a continuous basis in combination with docetaxel
  Other Names: PRMT5 inhibitor
  Arms: Non small cell lung cancer PF-06939999 plus docetaxel; Non small cell lung cancer dose finding

SUMMARY:
This is a Phase 1, open label, multi center, dose escalation and expansion, safety, tolerability, PK, and pharmacodynamics study of PF 06939999 in previously treated patients with advanced or metastatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced or metastatic NSCLC, urothelial carcinoma or HNSCC
* Progressed after at least 1 line of treatment and no more than 3 lines of treatment
* At least one measurable lesion as defined by RECIST version 1.1
* ECOG Performance Status 0 or 1
* Adequate Bone Marrow Function
* Adequate Renal Function
* Adequate Liver Function
* Resolved acute effects of any prior therapy

Exclusion Criteria:

* Known active uncontrolled or symptomatic CNS metastases.
* Major surgery, radiation therapy, systemic anti-cancer therapy or investigational drug(s) within 4 weeks prior to study entry.
* Active, uncontrolled infection, including COVID-19
* Known or suspected hypersensitivity to PF-06939999
* Inability to consume or absorb study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2022-04-27 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- United States (22):
  - Scottsdale Healthcare Hospitals d/b/a HonorHealth, Scottsdale, Arizona
  - Virginia G. Piper Cancer Pharmacy, Scottsdale, Arizona
  - Keck Hospital of USC, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Keck Medical Center of USC Pasadena, Pasadena, California
  - AdventHealth Celebration Infusion Center, Celebration, Florida
  - AdventHealth Medical Group Oncology Research at Celebration, Celebration, Florida
  - University Of Miami Hospital and Clinics/Sylvester Comprehensive Cancer Center, Miami, Florida
  - AdventHealth Orlando - Investigational Drug Services, Orlando, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - AdventHealth Orlando, Orlando, Florida
  - St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - St. Joseph Mercy Brighton, Brighton, Michigan
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Oncology IDS Pharmacy, Nashville, Tennessee
  - The University of Texas, Houston, Texas
  - NEXT Oncology, San Antonio, Texas
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Seattle Cancer Care Alliance, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Guo C, Liao KH, Li M, Wang IM, Shaik N, Yin D. PK/PD model-informed dose selection for oncology phase I expansion: Case study based on PF-06939999, a PRMT5 inhibitor. CPT Pharmacometrics Syst Pharmacol. 2023 Nov;12(11):1619-1625. doi: 10.1002/psp4.12882. Epub 2022 Nov 16. PMID 36394153
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3851001

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-eight participants were enrolled in the dose escalation part (Part 1A) and a 26 participants were enrolled in the dose expansion part (Part 2A, Part 2B and Part 2C). A total of 54 participants were assigned to treatment and treated. The study was terminated during dose expansion part due to strategy reason but not safety concerns. No enrollments occurred in Part 1B and Part 2D prior to study termination. In Part 2B, no enrollments occurred for the food-effect substudy.
Groups:
- Part 1A: PF-06939999 0.5 mg Once Daily (QD): Part 1 is dose escalation part. Participants received PF-06939999 0.5 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 0.5 mg Twice Daily (BID): Participants received PF-06939999 0.5 mg BID in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 1 mg BID: Participants received PF-06939999 1 mg BID in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 2 mg BID: Participants received PF-06939999 2 mg BID in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 4 mg BID: Participants received PF-06939999 4 mg BID in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 6 mg BID: Participants received PF-06939999 6 mg BID in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 8 mg QD: Participants received PF-06939999 8 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 6 mg QD: Participants received PF-06939999 6 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 4 mg QD: Participants received PF-06939999 4 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD: Part 2 is dose expansion part. Participants with NSCLC who had progressed after at least 1 line of checkpoint inhibitors and 1 line of platinum based chemotherapy (2L+) received PF-06939999 6 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD: Participants with urothelial carcinoma who had progressed after at least 1 line of standard of care systemic chemotherapy (cisplatin/carboplatin+ Gemcitabine; or methotrexate/vinblastine sulfate/doxorubicin hydrochloride/cisplatin [MVAC]) and checkpoint inhibitor (2L+) received PF-06939999 6 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD: Participants with HNSCC who had progressed after at least 1 line of standard of care systemic chemotherapy and 1 line of checkpoint inhibitor (2L+) received PF-06939999 6 mg QD in 28-day cycles up to 2 years or until disease progression.
Period: Overall Study
Arm/Group | Part 1A: PF-06939999 0.5 mg Once Daily (QD) | Part 1A: PF-06939999 0.5 mg Twice Daily (BID) | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Started | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5 | 14 | 2 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5 | 14 | 2 | 10
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 3 | 0 | 1
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1
Not completed — Progressive disease | 1 | 1 | 1 | 2 | 3 | 1 | 2 | 5 | 2 | 5 | 1 | 6
Not completed — Study terminated by sponsor | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Disease relapse | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Global deterioration of health status | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Refused further treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline analysis population included all enrolled participants who received at least 1 dose of study treatment.
Groups:
- Part 1A: PF-06939999 0.5 mg QD: Part 1 is dose escalation part. Participants received PF-06939999 0.5 mg QD in 28-day cycles up to 2 years or until disease progression.
- Part 1A: PF-06939999 0.5 mg BID: Participants received PF-06939999 0.5 mg BID in 28-day cycles up to 2 years or until disease progression.
- Total: Total of all reporting groups
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD | Total
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5 | 14 | 2 | 10 | 54
Age, Continuous [Mean (Standard Deviation); unit: Years] | 81.00 | 54.00 | 65.00 (5.66) | 57.67 (3.06) | 63.00 (16.46) | 57.25 (14.59) | 67.33 (6.66) | 54.83 (11.81) | 67.80 (12.38) | 64.86 (8.88) | 65.00 (7.07) | 65.70 (10.22) | 63.35 (10.61)
Age, Continuous [Median (Full Range); unit: Years] | 81.00 [81 to 81] | 54.00 [54 to 54] | 65.00 [61 to 69] | 57.00 [55 to 61] | 72.00 [44 to 73] | 59.50 [38 to 72] | 69.00 [60 to 73] | 59.00 [32 to 64] | 69.00 [50 to 84] | 66.50 [48 to 79] | 65.00 [60 to 70] | 67.50 [45 to 77] | 64.00 [32 to 84]
Age, Customized [Count of Participants; unit: Participants]
  <18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 3
  45-64 years | 0 | 1 | 1 | 3 | 0 | 2 | 1 | 5 | 2 | 6 | 1 | 3 | 25
  >=65 years | 1 | 0 | 1 | 0 | 2 | 1 | 2 | 0 | 3 | 8 | 1 | 7 | 26
  Unspecified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 3 | 3 | 7 | 1 | 0 | 23
  Male | 0 | 0 | 1 | 2 | 2 | 2 | 1 | 3 | 2 | 7 | 1 | 10 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 1 | 1 | 0 | 2 | 1 | 1 | 0 | 2 | 1 | 3 | 12
  Not Hispanic or Latino | 1 | 1 | 1 | 2 | 3 | 2 | 2 | 5 | 5 | 9 | 1 | 7 | 39
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 4
  White | 1 | 0 | 2 | 3 | 2 | 4 | 2 | 6 | 5 | 10 | 0 | 9 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Part 1A: Number of Participants With Dose-Limiting Toxicities (DLT)
Description: DLTs=any of the following adverse events (AEs) occurring in the DLT observation period (first treatment cycle):1) Any Grade 4 hematologic AEs; Grade 4 neutropenia, febrile neutropenia, Grade 3 neutropenia with infection, Grade 3 thrombocytopenia with ≥Grade 2 clinically significant bleeding, Grade 3 anemia requiring blood transfusion; 2) Any Grade ≥3 non-hematologic AEs; Grade 3 nausea/vomiting or diarrhea lasting ≥4 days after treatment, confirmed drug induced liver injury meeting Hy's law criteria; a hepatic transaminase or alkaline phosphatase level >10 times the upper limit of normal for participants with Grade 2 hepatic transaminase or alkaline phosphatase levels at baseline as a result of liver/bone metastasis; clinically important or persistent toxicities; 3) Any toxicity causing >2 weeks of dose delay; 4) any dose reduction due to AE during the first cycle. Grades of AEs were defined by National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0.
Time Frame: Baseline through day 29.
Population: The analysis population included participants in Part 1A who had at least one dose of study treatment and either experienced DLT or did not have major treatment deviations during the DLT observation period.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 2 | 3 | 6 | 4
Participants | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0

2. Primary Outcome: Part 1A: Number of Participants With Treatment-Emergent Adverse Events (TEAE)
Description: An AE was any untoward medical occurrence in a participant who received study treatment without regard to possibility of causal relationship. A serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Grades of AEs were defined by NCI CTCAE version 5.0. Grade 3 events = unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 events = events that caused participant to be in imminent danger of death. Grade 5 events = death related to an AE.
Time Frame: Baseline up to a minimum of 28 days after last dose of study treatment (maximum of 13 months)
Population: The analysis set included all participants in Part 1A who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5
Participants
  All-Causality TEAEs | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5
  All-Causality SAEs | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2 | 2
  Maximum Grade 3 or 4 All-Causality AEs | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 4 | 1
  Maximum Grade 5 All-Causality AEs | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1
  All-causality TEAEs Leading to Discontinuation From Study | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
  Treatment-related TEAEs | 1 | 1 | 1 | 2 | 3 | 2 | 3 | 6 | 5
  Treatment-related SAEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Maximum Grade 3 or 4 Treatment-related AEs | 0 | 0 | 1 | 1 | 2 | 2 | 2 | 2 | 2
  Maximum Grade 5 Treatment-related AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Treatment-related TEAEs leading to discontinuation form study | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Part 1A: Number of Participants With Laboratory Abnormalities
Description: Laboratory assessments included hematology, chemistry and urinary tests. Participants with maximum Grade 3-4 laboratory abnormalities are reported in this OM. Grades of laboratory results were defined by NCI CTCAE version 5.0. Grade 3 events = unacceptable or intolerable events, significantly interrupting usual daily activity, require systemic drug therapy/other treatment. Grade 4 events = events that caused participant to be in imminent danger of death. Some of the Grade 4 events (activated partial thromboplastin time prolonged, anemia, hemoglobin increased, leukocytosis, lymphocyte count increased and hypoalbuminemia) could not be defined/determined based only on lab data, therefore are not reported in this OM.
Time Frame: Baseline up to a minimum of 28 days after last dose of study treatment (maximum of 12 months)
Population: The analysis set included all participants in Part 1A who received at least 1 dose of study treatment. Number of Participants Analyzed = number of participants evaluable for this outcome measure. Number Analyzed = number of participants evaluable for the specific laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5
Participants
  Activated Partial Thromboplastin Time Prolonged (Grade 3): number analyzed (Participants) | 1 | 1 | 1 | 2 | 3 | 3 | 2 | 6 | 4
  Activated Partial Thromboplastin Time Prolonged (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Anemia (Grade 3) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 2 | 2
  Hemoglobin Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytosis (Grade 3): number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 4 | 3 | 6 | 5
  Leukocytosis (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Decreased (Grade 3) | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 3 | 2
  Lymphocyte Count Decreased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocyte Count Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Neutrophil Count Decreased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Neutrophil Count Decreased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Platelet Count Decreased (Grade 3) | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0
  Platelet Count Decreased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  White Blood Cell Decreased (Grade 3): number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 4 | 3 | 6 | 5
  White Blood Cell Decreased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White Blood Cell Decreased (Grade 4): number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 4 | 3 | 6 | 5
  White Blood Cell Decreased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alanine Aminotransferase Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Alanine Aminotransferase Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Alkaline Phosphatase Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Aspartate Aminotransferase Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
  Aspartate Aminotransferase Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Creatinine Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Creatinine Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypercalcemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hyperkalemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypermagnesemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypernatremia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoalbuminemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Hypocalcemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypocalcemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypoglycemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypokalemia (Grade 3) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
  Hypokalemia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Hypomagnesemia (Grade 4) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Hyponatremia (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Hyponatremia (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Lipase Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serum Amylase Increased (Grade 3) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Serum Amylase Increased (Grade 4) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Part 2: Number of Participants With TEAEs
Description: as for outcome 2
Time Frame: Baseline up to a minimum of 28 days after last dose of study treatment (maximum of 15 months)
Population: The analysis set included all participants in Part 2 who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 14 | 2 | 10
Participants
  All-Causality TEAEs | 14 | 2 | 10
  All-Causality SAEs | 7 | 1 | 5
  Maximum Grade 3 or 4 All-Causality AEs | 11 | 2 | 5
  Maximum Grade 5 All-Causality AEs | 3 | 0 | 2
  All-causality TEAEs Leading to Discontinuation From Study | 3 | 0 | 2
  Treatment-related TEAEs | 10 | 2 | 9
  Treatment related SAEs | 1 | 1 | 1
  Maximum Grade 3 or 4 Treatment-related AEs | 5 | 2 | 4
  Maximum Grade 5 Treatment-related AEs | 0 | 0 | 0
  Treatment-related TEAEs leading to discontinuation form study | 0 | 0 | 0

5. Primary Outcome: Part 2: Number of Participants With Laboratory Abnormalities
Description: as for outcome 3
Time Frame: Baseline up to a minimum of 28 days after last dose of study treatment (maximum of 8 months)
Population: The analysis set included all participants in Part 2 who received at least 1 dose of study treatment. Number of Participants Analyzed = number of participants evaluable for this outcome measure. Number Analyzed = number of participants evaluable for the specific laboratory test.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 14 | 2 | 10
Participants
  Activated Partial Thromboplastin Time Prolonged (Grade 3): number analyzed (Participants) | 11 | 2 | 8
  Activated Partial Thromboplastin Time Prolonged (Grade 3) | 1 | 0 | 1
  Anemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Anemia (Grade 3) | 5 | 1 | 2
  Hemoglobin Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hemoglobin Increased (Grade 3) | 0 | 0 | 0
  Leukocytosis (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Leukocytosis (Grade 3) | 0 | 0 | 0
  Lymphocyte Count Decreased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Lymphocyte Count Decreased (Grade 3) | 4 | 1 | 3
  Lymphocyte Count Decreased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Lymphocyte Count Decreased (Grade 4) | 0 | 0 | 3
  Lymphocyte Count Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Lymphocyte Count Increased (Grade 3) | 0 | 0 | 0
  Neutrophil Count Decreased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Neutrophil Count Decreased (Grade 3) | 1 | 0 | 0
  Neutrophil Count Decreased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Neutrophil Count Decreased (Grade 4) | 0 | 0 | 0
  Platelet Count Decreased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Platelet Count Decreased (Grade 3) | 2 | 1 | 2
  Platelet Count Decreased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Platelet Count Decreased (Grade 4) | 1 | 0 | 0
  White Blood Cell Decreased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  White Blood Cell Decreased (Grade 3) | 1 | 0 | 0
  White Blood Cell Decreased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  White Blood Cell Decreased (Grade 4) | 0 | 0 | 0
  Alanine Aminotransferase Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Alanine Aminotransferase Increased (Grade 3) | 0 | 0 | 0
  Alanine Aminotransferase Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Alanine Aminotransferase Increased (Grade 4) | 0 | 0 | 0
  Alkaline Phosphatase Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Alkaline Phosphatase Increased (Grade 3) | 0 | 0 | 0
  Alkaline Phosphatase Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Alkaline Phosphatase Increased (Grade 4) | 0 | 0 | 0
  Aspartate Aminotransferase Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Aspartate Aminotransferase Increased (Grade 3) | 0 | 0 | 0
  Aspartate Aminotransferase Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Aspartate Aminotransferase Increased (Grade 4) | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Blood Bilirubin Increased (Grade 3) | 0 | 0 | 0
  Blood Bilirubin Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Blood Bilirubin Increased (Grade 4) | 0 | 0 | 0
  Creatinine Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Creatinine Increased (Grade 3) | 0 | 0 | 0
  Creatinine Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Creatinine Increased (Grade 4) | 1 | 0 | 0
  Hypercalcemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypercalcemia (Grade 3) | 0 | 0 | 1
  Hypercalcemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypercalcemia (Grade 4) | 1 | 0 | 0
  Hyperkalemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hyperkalemia (Grade 3) | 0 | 0 | 0
  Hyperkalemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hyperkalemia (Grade 4) | 0 | 0 | 0
  Hypermagnesemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypermagnesemia (Grade 3) | 0 | 0 | 0
  Hypermagnesemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypermagnesemia (Grade 4) | 0 | 0 | 0
  Hypernatremia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypernatremia (Grade 3) | 0 | 0 | 0
  Hypernatremia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypernatremia (Grade 4) | 0 | 0 | 0
  Hypoalbuminemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypoalbuminemia (Grade 3) | 0 | 0 | 0
  Hypocalcemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypocalcemia (Grade 3) | 0 | 0 | 0
  Hypocalcemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypocalcemia (Grade 4) | 0 | 0 | 0
  Hypoglycemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypoglycemia (Grade 3) | 0 | 0 | 0
  Hypoglycemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypoglycemia (Grade 4) | 0 | 0 | 0
  Hypokalemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypokalemia (Grade 3) | 1 | 0 | 1
  Hypokalemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypokalemia (Grade 4) | 0 | 0 | 0
  Hypomagnesemia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hypomagnesemia (Grade 3) | 0 | 0 | 0
  Hypomagnesemia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hypomagnesemia (Grade 4) | 0 | 0 | 0
  Hyponatremia (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Hyponatremia (Grade 3) | 1 | 1 | 2
  Hyponatremia (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Hyponatremia (Grade 4) | 0 | 0 | 0
  Lipase Increased (Grade 3): number analyzed (Participants) | 11 | 2 | 10
  Lipase Increased (Grade 3) | 0 | 0 | 0
  Lipase Increased (Grade 4): number analyzed (Participants) | 11 | 2 | 10
  Lipase Increased (Grade 4) | 0 | 0 | 0
  Serum Amylase Increased (Grade 3): number analyzed (Participants) | 13 | 2 | 10
  Serum Amylase Increased (Grade 3) | 0 | 0 | 0
  Serum Amylase Increased (Grade 4): number analyzed (Participants) | 13 | 2 | 10
  Serum Amylase Increased (Grade 4) | 0 | 0 | 0

6. Primary Outcome: Part 2: Number of Participants With Best Overall Response (BOR) Based on Investigator Assessment (RECIST, Version 1.1)
Description: Number of participants with BOR assessed using Response Evaluation Criteria in Solid Tumor (RECIST) v1.1: Complete Response (CR): disappearance of all lesions (with the exception of nodal disease when assessing target lesions). Partial Response (PR): at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters. Progressive Disease (PD): at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered a sign of progression. Stable disease (SD): does not qualify for CR, PR or PD. Non-CR/Non-PD: Persistence of any non target lesions and/or tumor marker level above the normal limits.
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 6 months).
Population: The analysis population included all participants in Part 2 who received at least one dose of study treatment and had baseline disease assessment or measurable disease at baseline, if applicable and at least one post baseline disease assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 11 | 2 | 8
Participants
  Complete response (CR) | 0 | 0 | 0
  Partial response (PR) | 1 | 0 | 0
  Stable disease (SD) | 4 | 2 | 4
  Non-CR/Non-PD | 0 | 0 | 0
  Progressive disease (PD) | 4 | 0 | 4
  Not evaluable (NE) | 2 | 0 | 0

7. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: Single Dose (SD) - Maximum Observed Plasma Concentration (Cmax)
Description: Maximum plasma concentration of PF-06939999 after the participant received a SD on Cycle 1 Day 1. Cmax was directly observed from data.
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours, 4 hours, 6 hours and 12 hours post the morning dose on Cycle 1 Day 1.
Population: The analysis population included enrolled participants in Part 1A treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5
nanogram per milliliter (ng/mL) | NA (NA) — Geometric mean and geometric coefficient of variation (CV) are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 6.295 (13) | 26.33 (70) | 26.64 (63) | 52.96 (85) | 28.56 (72) | 21.63 (82)

8. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: SD - Time to Reach Maximum Observed Plasma Concentration (Tmax)
Description: Time to maximum plasma concentration of PF-06939999 after the participant received a SD on Cycle 1 Day 1. Tmax was observed directly from data.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 1.
Population: as for outcome 7
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 3 | 3 | 4 | 3 | 6 | 5
hours (hr) | 0.9 [0.9 to 0.9] | 2.0 [2.0 to 2.0] | 2.1 [2.1 to 2.1] | 1.0 [0.5 to 2.1] | 1.0 [0.5 to 3.7] | 1.5 [0.5 to 4.0] | 2.0 [1.0 to 2.1] | 1.5 [0.7 to 2.2] | 0.9 [0.5 to 4.3]

9. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: SD - Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration versus time curve (AUC) from time 0 to the last measured concentration (AUClast) after the participant received a SD of PF-06939999 on Cycle 1 Day 1.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 1.
Population: The analysis population included enrolled participants in Part 1A treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest with evaluable data that contributed to the summary statistics of this outcome measure (OM).
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram*hour per milliliter (ng*hr/mL)
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 0 | 0 | 2 | 3 | 3 | 4 | 2 | 4 | 4
nanogram*hour per milliliter (ng*hr/mL) |  |  | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 20.52 (15) | 93.77 (61) | 88.94 (51) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 256.7 (75) | 136.4 (94)

10. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: Multiple Dose (MD) - Steady State Maximum Observed Plasma Concentration (Cmax,ss)
Description: Cmax,ss was the steady-state maximum concentration of PF-06939999 after MD. Cmax,ss was observed directly from the data.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 15.
Population: The analysis population included enrolled participants in Part 1A treated who did not had protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest, with evaluable data that contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 6 | 3
ng/mL | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 59.78 (37) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 59.32 (26) | 29.39 (99)

11. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: MD - Steady State Time to Reach Maximum Observed Plasma Concentration (Tmax,ss)
Description: Tmax,ss was the steady-state time to maximum plasma concentration of PF-06939999 after MD. Tmax,ss was observed directly from data.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 15.
Population: The analysis population included enrolled participants in Part 1A treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest, with evaluable data that contributed to the summary statistics of this OM.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 6 | 3
hr | 0.5 [0.5 to 0.5] | 5.6 [5.6 to 5.6] | 0.75 [0.5 to 1.0] | 1.6 [1.0 to 2.2] | 0.5 [0.5 to 1.9] | 1.0 [1.0 to 1.0] | 1.5 [1.0 to 2.0] | 1.0 [0.5 to 2.2] | 1.9 [0.5 to 2.1]

12. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: MD - Area Under the Curve From Time Zero to End of Dosing Interval (AUCtau,ss)
Description: AUCtau,ss was the steady-state area under the concentration-time profile from time zero to time tau (τ) of PF-06939999 after MD.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 15.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 6 | 3
ng*hr/mL | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 437.4 (31) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 718.3 (38) | 360.6 (98)

13. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: MD - Apparent Oral Clearance (CL/F)
Description: Apparent oral plasma clearance of PF-06939999 after MD. CL/F after multiple doses = Dose/AUCtau,ss. AUCtau,ss = area under the concentration-time profile from time zero to time tau after multiple doses.
Time Frame: Predose, 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 15.
Population: as for outcome 11
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour (L/hr)
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 1 | 2 | 6 | 3
liters per hour (L/hr) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 9.163 (31) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 8.358 (38) | 11.09 (98)

14. Secondary Outcome: Part 1A: PK Parameters of PF-06939999: MD - Accumulation Ratio (Rac)
Description: Rac was observed accumulation ratio based on AUCtau. Rac was calculated as AUCtau (multiple dose, Cycle 1 Day 15)/ AUCtau (single dose, Cycle 1 Day 1). AUCtau was area under the concentration-time profile from time zero to time tau (τ), the dosing interval.
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours, 4 hours, 6 hours and 12 hours post the morning dose on Cycle 1 Day 1; Pre-dose and 0.5, 1, 2, 4, 6 and 12 hours post the morning dose on Cycle 1 Day 15.
Population: The analysis population included enrolled participants in Part 1A treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest, and contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 0 | 0 | 2 | 2 | 2 | 1 | 1 | 4 | 3
ratio |  |  | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 3.262 (52) | 2.526 (20)

15. Secondary Outcome: Part 2: PK Parameters of PF-06939999: SD - Cmax
Description: as for outcome 7
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours and 4 hours post Cycle 1 Day 1 dosing.
Population: The analysis population included enrolled participants in Part 2 treated who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest, with evaluable data that contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 13 | 2 | 10
ng/mL | 38.60 (93) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 30.89 (50)

16. Secondary Outcome: Part 2: PK Parameters of PF-06939999: SD - Tmax
Description: as for outcome 8
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours and 4 hours post Cycle 1 Day 1 dosing.
Population: as for outcome 15
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 13 | 2 | 10
hr | 0.9 [0.5 to 2.2] | 1.25 [0.5 to 2.0] | 1.0 [0.9 to 2.0]

17. Secondary Outcome: Part 2: PK Parameters of PF-06939999: MD - Cmax,ss
Description: Cmax,ss was the steady-state maximum concentration of PF-06939999 after MD. Cmax,ss was observed directly from the data.
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours and 4 hours post Cycle 1 Day 15 dosing.
Population: The analysis population included enrolled participants in Part 2 treated who did not have protocol deviations influencing PK assessment, and have sufficient information to estimate at least 1 of the PK parameters of interest, with evaluable data that contributed to the summary statistics of this OM.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 9 | 2 | 7
ng/mL | 81.27 (57) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 50.22 (40)

18. Secondary Outcome: Part 2: PK Parameters of PF-06939999: MD - Tmax,ss
Description: as for outcome 11
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours and 4 hours post Cycle 1 Day 15 dosing.
Population: as for outcome 17
Measure: Median (Full Range); unit: hr
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 9 | 2 | 7
hr | 1.1 [0.5 to 4.0] | 2.05 [2.0 to 2.1] | 2.1 [1.0 to 4.0]

19. Secondary Outcome: Part 2: PK Parameters of PF-06939999: MD - Trough Concentration (Ctrough).
Description: Ctrough was trough serum concentration of PF-06939999 after MD. Ctrough = Cmin.
Time Frame: Pre-dose and 0.5 hour, 1 hour, 2 hours and 4 hours post Cycle 1 Day 15 dosing.
Population: as for outcome 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 9 | 2 | 7
ng/mL | 21.55 (93) | NA (NA) — Geometric mean and geometric CV are not applicable due to n<3. | 17.33 (61)

20. Secondary Outcome: Part 2B: PK Parameters of PF-06939999 Given With and Without Food - Cmax
Description: Maximum concentration of PF-06939999 given with and without food. On Cycle 1 Day 15, participants enrolled in the food-effect substudy of Part 2B received an oral dose of PF-06939999 under the fasted condition (overnight fasting of at least 10 hours; water permitted). On Cycle 1 Day 16, these participants received another oral dose of PF-06939999 with a high-fat, high-calorie meal (breakfast) following 10-hour overnight fasting (water permitted).
Time Frame: Predose and 0.5, 1, 2, 4, 6 and 12 hours post dose on Cycle 1 Day 15 (fasted condition); predose and 0.5, 1, 2, 4, 6 and 12 hours post dose on Cycle 1 Day 16 (with food).
Population: The analysis population included participants enrolled and treated in the food-effect substudy of Part 2B who did not have protocol deviations influencing PK assessment, and had sufficient information to estimate at least 1 of the PK parameters of interest. Food-effect cohort in Part 2B was not enrolled.
Arm/Group | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD
Number analyzed (Participants) | 0

21. Secondary Outcome: Part 2B: PK Parameters of PF-06939999 Given With and Without Food - Tmax
Description: Time to maximum plasma concentration of PF-06939999 given with and without food. On Cycle 1 Day 15, participants enrolled in the food-effect substudy of Part 2B received an oral dose of PF-06939999 under the fasted condition (overnight fasting of at least 10 hours; water permitted). On Cycle 1 Day 16, these participants received another oral dose of PF-06939999 with a high-fat, high-calorie meal (breakfast) following 10-hour overnight fasting (water permitted).
Time Frame: as for outcome 20
Population: as for outcome 20
Arm/Group | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD
Number analyzed (Participants) | 0

22. Secondary Outcome: Part 2B: PK Parameters of PF-06939999 Given With and Without Food - AUClast
Description: AUClast of PF-06939999 given with and without food. On Cycle 1 Day 15, participants enrolled in the food-effect substudy of Part 2B received an oral dose of PF-06939999 under the fasted condition (overnight fasting of at least 10 hours; water permitted). On Cycle 1 Day 16, these participants received another oral dose of PF-06939999 with a high-fat, high-calorie meal (breakfast) following 10-hour overnight fasting (water permitted).
Time Frame: as for outcome 20
Population: as for outcome 20
Arm/Group | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD
Number analyzed (Participants) | 0

23. Secondary Outcome: Part 1A: Percentage of Participants With Objective Response Based on Investigator Assessment (RECIST v1.1)
Description: Objective Response Rate (ORR) was defined as the percentage of participants who achieved CR or PR per RECIST 1.1. CR was defined as disappearance of all lesions. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 12 months).
Population: The analysis population included all participants in Part 1A who received at least one dose of study treatment and had baseline disease assessment or measurable disease at baseline, if applicable and at least one post baseline disease assessment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 1 | 1 | 2 | 2 | 3 | 2 | 2 | 6 | 4
Percentage of participants | 0 [0.0 to 79.3] | 0 [0.0 to 79.3] | 0 [0.0 to 65.8] | 50.0 [9.5 to 90.5] | 33.3 [6.1 to 79.2] | 0 [0.0 to 65.8] | 0 [0.0 to 65.8] | 0 [0.0 to 39.0] | 0 [0.0 to 49.0]

24. Secondary Outcome: Part 1A: Duration of Response Based on Investigator Assessment (RECIST, v1.1)
Description: Duration of response was defined as the time from start date (which is the date of first documentation of PR or CR) to date of first documentation of objective progression or death. DOR was only applicable to those participants with an objective response (confirmed CR or PR). CR: disappearance of all lesions (with the exception of nodal disease when assessing target lesions). PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 12 months).
Population: The analysis population included all participants in Part 1A who received at least one dose of study treatment and had baseline disease assessment or measurable disease at baseline, if applicable and at least one post baseline disease assessment, with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD
Number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Months |  |  |  | 4.3 [NA to NA] — 95% Confidence Interval (CI) is not applicable due to n = 1. | 4.7 [NA to NA] — 95% CI is not applicable due to n = 1. |  |  |  |

25. Secondary Outcome: Part 2: Duration of Response Based on Investigator Assessment (RECIST, v1.1)
Description: as for outcome 24
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 6 months).
Population: The analysis population included all participants in Part 2 who received at least one dose of study treatment and had baseline disease assessment or measurable disease at baseline, if applicable and at least one post baseline disease assessment, with confirmed CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 1 | 0 | 0
Months | NA [NA to NA] — Median and 95% CI are not applicable due to insufficient number of participants with events. |  |

26. Secondary Outcome: Part 2: Progression Free Survival Based on Investigator Assessment (RECIST, v1.1)
Description: Progression Free Survival (PFS) was defined as the time from initiation of PF-06939999 therapy to first documentation of tumor progression or to death due to any cause, whichever occurred first.
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 6 months).
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 11 | 2 | 8
Months | 3.4 [1.1 to NA] — The upper limit of 95% CI is not applicable due to insufficient number of participants with events. | 5.5 [NA to NA] — 95% CI is not applicable due to insufficient number of participants with events. | 1.9 [1.6 to 5.6]

27. Secondary Outcome: Part 2: Time to Progression Based on Investigator Assessment (RECIST, v1.1)
Description: Time to Progression (TTP) was defined as the time from the date of the first treatment to the date of the first documentation of objective tumor progression or death due to tumor progression. Disease progression is defined using RECIST v 1.1.
Time Frame: From baseline up to 28 ~ 35 days after end of treatment (maximum of 6 months).
Population: as for outcome 6
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 11 | 2 | 8
Months | 3.4 [1.1 to NA] — The upper limit of 95% CI is not applicable due to insufficient number of participants with events. | 5.5 [NA to NA] — 95% CI is not applicable due to insufficient number of participants with events. | 1.9 [1.6 to 5.6]

28. Secondary Outcome: Part 2: Overall Survival
Description: Overall Survival (OS) was defined as the time from the start date (first dose) of study treatment to the date of death due to any cause.
Time Frame: From baseline up to maximum follow up (15 months).
Population: The analysis set included all participants in Part 2 who received at least 1 dose of study treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 14 | 2 | 10
Months | 6.0 [1.0 to NA] — The upper limit of 95% CI is not applicable due to insufficient number of participants with events. | NA [NA to NA] — Median and 95% CI are not applicable due to insufficient number of participants with events. | 14.6 [0.8 to NA] — The upper limit of 95% CI is not applicable due to insufficient number of participants with events.

29. Secondary Outcome: Part 2: Probability of Survival at 6 Months and 1 Year of PF-06939999 Monotherapy
Description: The probability of survival at select times was estimated using the Kaplan Meier method. Although an endpoint of Overall Survival at 2 years of study treatment was defined in the protocol, no data were collected/analyzed for this endpoint due to maximum follow up not reaching 2 year post study treatment.
Time Frame: From baseline up to maximum follow up (15 months).
Population: The analysis set included all participants in Part 2 who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: probability of survival
Arm/Group | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
Number analyzed (Participants) | 14 | 2 | 10
probability of survival
  6 Months | 0.550 [0.258 to 0.768] | 1.000 [1.000 to 1.000] | 0.778 [0.365 to 0.939]
  1 Year | 0.283 [0.073 to 0.543] | NA [NA to NA] — Probability of survival and 95% CI are not applicable due to insufficient number of participants with events. | 0.519 [0.084 to 0.840]

ADVERSE EVENTS:
Time Frame: Baseline up to a minimum of 28 days after last dose of study treatment (part 1 maximum of 13 months, part 2 maximum of 15 months)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study.
Arm/Group | Part 1A: PF-06939999 0.5 mg QD | Part 1A: PF-06939999 0.5 mg BID | Part 1A: PF-06939999 1 mg BID | Part 1A: PF-06939999 2 mg BID | Part 1A: PF-06939999 4 mg BID | Part 1A: PF-06939999 6 mg BID | Part 1A: PF-06939999 8 mg QD | Part 1A: PF-06939999 6 mg QD | Part 1A: PF-06939999 4 mg QD | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 0/3 | 0/3 | 2/4 | 1/3 | 0/6 | 1/5 | 9/14 | 0/2 | 4/10
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/2 | 1/3 | 0/3 | 3/4 | 1/3 | 2/6 | 2/5 | 7/14 | 1/2 | 5/10
Other Adverse Events (participants affected / at risk) | 1/1 | 1/1 | 2/2 | 3/3 | 3/3 | 4/4 | 3/3 | 6/6 | 5/5 | 12/14 | 2/2 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: PF-06939999 0.5 mg QD (N=1) | Part 1A: PF-06939999 0.5 mg BID (N=1) | Part 1A: PF-06939999 1 mg BID (N=2) | Part 1A: PF-06939999 2 mg BID (N=3) | Part 1A: PF-06939999 4 mg BID (N=3) | Part 1A: PF-06939999 6 mg BID (N=4) | Part 1A: PF-06939999 8 mg QD (N=3) | Part 1A: PF-06939999 6 mg QD (N=6) | Part 1A: PF-06939999 4 mg QD (N=5) | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD (N=14) | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD (N=2) | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 2 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Radiation necrosis (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Arterial rupture (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: PF-06939999 0.5 mg QD (N=1) | Part 1A: PF-06939999 0.5 mg BID (N=1) | Part 1A: PF-06939999 1 mg BID (N=2) | Part 1A: PF-06939999 2 mg BID (N=3) | Part 1A: PF-06939999 4 mg BID (N=3) | Part 1A: PF-06939999 6 mg BID (N=4) | Part 1A: PF-06939999 8 mg QD (N=3) | Part 1A: PF-06939999 6 mg QD (N=6) | Part 1A: PF-06939999 4 mg QD (N=5) | Part 2A: [2L+ Non-small Cell Lung Cancer (NSCLC)] PF-06939999 6mg QD (N=14) | Part 2B: (2L+ Urothelial Carcinoma) PF-06939999 6mg QD (N=2) | Part 2C: [2L+ Head and Neck Squamous Cell Carcinoma (HNSCC)] PF-06939999 6mg QD (N=10)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 3 | 4 | 1 | 5
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 2 | 2 | 2 | 1 | 1 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scleral oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anal incontinence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 3 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 0 | 2 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2 | 1 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 5 | 2 | 7 | 0 | 4
Pancreatic failure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 2 | 0 | 3 | 0 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 2 | 2 | 1 | 1 | 4 | 3 | 4 | 0 | 5
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Skin candida (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Soft tissue infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Animal scratch (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lipase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 1 | 2
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 3
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 1 | 5 | 0 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 5 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Brain oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 3 | 1 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device malfunction (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Irritability (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nephropathy (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 2 | 1 | 0 | 0 | 1 | 2 | 1 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Orthostatic hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
The study was terminated based on a strategic decision. This decision was not due to any safety concerns or requests from any regulatory authorities.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-06-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT03854227/Prot_000.pdf
  • Statistical Analysis Plan (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT03854227/SAP_001.pdf